CLINICAL TRIAL: NCT02557425
Title: Prophylaxis Against Malaria to Enhance Child Development
Brief Title: Prophylaxis Against Malaria to Enhance Child Development (PROTECT Study)
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Chandy John, Professor of Pediatrics, Indiana University
Other Study IDs: 1506994146
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Neurobehavioral Manifestations
Keywords: malaria; infant; pregnancy; prophylaxis; dihyroartemisinin-piperaquine; sulfadoxine-pyrimethamine; behavior; neurodevelopment; cognitive
MeSH Terms: conditions — Neurobehavioral Manifestations; Malaria; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Maternal SP/Child 3mo DP: In this group in the PROMOTE-II study, mothers receive 3 doses of sulfadoxine-pyrimethamine (SP), and children receive every 3 month dihydroartemisinin-piperaquine (DP). No intervention is given in the observational PROTECT study.
  Interventions: Other: No intervention in PROTECT
- Maternal 3 dose DP/Child 3mo DP: In this group in the PROMOTE-II study, mothers receive 3 doses of DP, and children receive every 3 month DP.No intervention is given in the observational PROTECT study.
  Interventions: Other: No intervention in PROTECT
- Maternal 3 dose DP/Child monthly DP: In this group in the PROMOTE-II study, mothers receive 3 doses of DP, and children receive monthly DP. No intervention is given in the observational PROTECT study.
  Interventions: Other: No intervention in PROTECT
- Maternal monthly DP/Child 3mo DP: In this group in the PROMOTE-II study, mothers receive monthly DP, and children receive every 3 month DP. No intervention is given in the observational PROTECT study.
  Interventions: Other: No intervention in PROTECT
- Maternal monthly DP/child monthly DP: In this group in the PROMOTE-II study, mothers receive monthly DP, and children receive every monthly DP. No intervention is given in the observational PROTECT study.
  Interventions: Other: No intervention in PROTECT

INTERVENTIONS:
Other: No intervention in PROTECT

SUMMARY:
Each year, ~85.3 million pregnant women are at risk of becoming infected with Plasmodium falciparum(1). Among women in sub-Saharan Africa, most of whom have some degree of clinical immunity to malaria, malaria infection in pregnancy leads to placental malaria (PM), often without clinical symptoms in the mother. The systemic and placental changes that occur with malaria in pregnancy can adversely affect the developing fetal brain, an fetal brain injury strongly affects long-term childhood neurodevelopmental (ND) and behavior but there are no published studies to date on the impact of malaria in pregnancy on childhood ND. This study, conducted in Uganda, will address the effects of malaria in pregnancy and childhood ND and define mechanisms by which malaria may lead to ND impairment including micronutrient deficiencies. ND outcomes will be measured by the following neuropsychological and behavioral tests: Mullen Scales of Early Learning, the Color Object Association Test, the Early Childhood Vigilance Test, the Behavior Rating Scales, the Behavior Related inventory of Executive Function and the Child Behavior Checklist. These tests will be given at 12, 24, 36, and 60 months of age. This study will be nested in an ongoing Ugandan IRB approved interventional trial (PROMOTE-II) (NCT02163447). Blood sampling is being conducted in the PROMOTE-II protocol for research purposes. Some of that blood will be used to test for micronutrient deficiencies as well as other immune responses to malaria.

DETAILED DESCRIPTION:
The PROMOTE-II randomized clinical trial in Tororo, Uganda, led by investigators from Makerere University in Uganda and the University of California-San Francisco (UCSF), provides an ideal setting to assess the effects of malaria prevention in pregnant women and their children on childhood ND. In PROMOTE-II Project 1,300 pregnant HIV-uninfected women will be randomized at 12-20 weeks of gestation to malaria prophylaxis with 3 doses of sulfadoxine-pyrimethamine (current standard of care), 3 doses of dihydroartemisinin-piperaquine (DP), or monthly DP. Their children will be randomized to receive DP prophylaxis monthly or every 3 months from 2 to 24 months age. The children will be followed for malaria episodes from birth to age 36 months. The proposed prospective study of child ND, the Prophylaxis against malaria To Enhance Child developmenT (PROTECT) study, will be nested within the PROMOTE-II Project 1 cohort. It is hypothesized that mothers on SP and mothers and children on less frequent prophylaxis will have more malaria episodes. The investigators predict that child ND will improve with more effective prophylaxis.

The central hypotheses of this study are that malaria prevention in pregnant women and their children improves child ND through 1) prevention of placental sequestration and inflammation and of consequent micronutrient deficiency in the fetus, and 2) reduction of systemic inflammation and endothelial activation that can lead to micronutrient deficiency and anemia during pregnancy and in early childhood and thus to alteration of brain structures particularly sensitive to such deficiencies (e.g., the hippocampus, myelin and the frontal lobe). The collaborative team, which has expertise in malaria in pregnant women and children, malaria pathogenesis, micronutrient deficiency, fetal and child neurodevelopment, and modeling of complex disease pathways, is well qualified to undertake the proposed research.

The specific aims of the study are:

Aim 1. Determine the effect of malaria prevention in pregnant women and their children on child ND. Hypotheses: 1) Long-term child ND improves with more effective chemoprevention in pregnant women and in their children. 2) The effect of malaria prevention on child ND persists through 36 months of age. Child ND will be assessed with a testing battery validated in previous studies by this group in Ugandan children. The investigators will test these hypotheses by comparing child ND at 12, 24, 36 and 60 months of age between treatment groups.

Aim 2. Identify the major mechanisms by which malaria prevention in pregnant women and children affects child ND. Hypotheses: 1) Malaria prevention in pregnant women affects child ND through prevention of placental sequestration and inflammation, with consequent prevention of prematurity, intrauterine growth retardation and fetal micronutrient deficiency. 2) Malaria prevention in pregnant women and in their children after birth improves child ND through reduction of systemic inflammation, endothelial activation, micronutrient deficiency and anemia, but the relative contributions of the factors differ in pregnant women compared to children. The investigators will test these hypotheses by conducting path analysis to determine if networks that include these paths explain a significant proportion of the difference in child ND between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in Makerere University-UCSF PROMOTE II study
2. HIV-uninfected
3. 12 months of age at the time of enrollment
4. Within 30 km of the clinic

Exclusion Criteria:

1. Serious adverse event to the study drugs requiring cessation of study drug
2. Active illness at enrollment (child can be enrolled once active illness has been treated and they are back to baseline health)
3. Previous history of head trauma or coma in the child
4. Cerebral palsy or other severe neurologic disease
5. Known chronic illness requiring medical care
6. Major medical abnormalities on screening history of past health
7. Known developmental delay

Ages: 10 Months to 38 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 300 Ugandan Children already enrolled in PROMOTE II study
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2015-10; Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Z-scores for Overall cognitive ability | 12 months of age
Z-scores for Overall cognitive ability | 24 months of age
Z-scores for Overall cognitive ability | 36 months of age
Z scores for Elicited Imitation | 12 months of age
Z scores for Elicited Imitation | 24 months of age
Z scores for Elicited Imitation | 36 months of age
Z scores of Overal Cognitive ability | 60 months of age
Z scores of Elicited Imitation | 60 months of age

SECONDARY OUTCOMES:
Z scores for Behavioral Rating Scale | 24, 36, and 60 months of age
Z scores for Behavior Related Inventory of Executive Function (BRIEF) | 24, 36, and 60 months of age
Z scores for Child Behavior Checklist (CBCL) | 24, 36, and 60 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C John, MD, Principal Investigator — Indiana University
Locations (1):
- Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Derived] Bangirana P, Conroy AL, Opoka RO, Semrud-Clikeman M, Jang JH, Apayi C, Kakuru A, Muhindo MK, Georgieff MK, Dorsey GM, Kamya MR, Havlir D, John CC. Effect of Malaria and Malaria Chemoprevention Regimens in Pregnancy and Childhood on Neurodevelopmental and Behavioral Outcomes in Children at 12, 24, and 36 Months: A Randomized Clinical Trial. Clin Infect Dis. 2023 Feb 18;76(4):600-608. doi: 10.1093/cid/ciac815. PMID 36219705